CLINICAL TRIAL: NCT00139945
Title: Effects of Acute Ghrelin Infusion to Growth Hormone Deficient Adults: Growth Hormone and Cortisol Interaction
Brief Title: Ghrelin, Growth Hormone and Cortisol Interaction in Growth Hormone Deficient Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Esben T. Vestergaard/MD PhD, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004/102
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Hypopituitarism
MeSH Terms: conditions — Hypopituitarism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Human acylated ghrelin — 5 pmol/kg body weight per min

SUMMARY:
In growth hormone deficient patients: Determination of endogenous circulating ghrelin levels, ghrelin effects on insulin sensitivity, appetite, energy metabolism, and signal transduction in fat and muscle.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 yrs.
* Verified hypopituitarism
* Unchanged substitution treatment through 3+ months
* Unchanged additional medical treatment
* Oral and written informed consent

Exclusion Criteria:

* Age below 18 or above 60 yrs.
* Diabetes mellitus
* body mass index > 30
* Fasting hypoglycemia
* Convulsions
* Allergy to trial products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Endogenous serum ghrelin levels | Same day as intervention

SECONDARY OUTCOMES:
Insulin sensitivity, appetite, metabolism, intracellular signal transduction | Same day as intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jorgensen, DrMedSci, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Lauritzen ES, Jorgensen JOL, Moller N, Nielsen S, Vestergaard ET. Increased lipolysis after infusion of acylated ghrelin: a randomized, double-blinded placebo-controlled trial in hypopituitary patients. Clin Endocrinol (Oxf). 2020 Dec;93(6):672-677. doi: 10.1111/cen.14290. Epub 2020 Aug 3. PMID 32975853
- [Derived] Vestergaard ET, Gormsen LC, Jessen N, Lund S, Hansen TK, Moller N, Jorgensen JO. Ghrelin infusion in humans induces acute insulin resistance and lipolysis independent of growth hormone signaling. Diabetes. 2008 Dec;57(12):3205-10. doi: 10.2337/db08-0025. Epub 2008 Sep 5. PMID 18776138